CLINICAL TRIAL: NCT00466167
Title: A Double-blind, Double-dummy, Placebo-controlled, Randomized, Three Parallel Groups Study Comparing the Efficacy, Safety and Tolerability of Pramipexole Extended Release (ER) Versus Placebo and Versus Pramipexole Immediate Release (IR) Administered Orally Over a 26-week Maintenance Phase in L-Dopa+ Treated Patients With Advanced Parkinsons Disease (PD).
Brief Title: Pivotal Study in Advanced Parkinsons Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: 248.525
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

ARMS (3):
- Pramipexole ER (Other)
  Interventions: Drug: Pramipexol Extended Release
- Pramipexole IR (Other)
  Interventions: Drug: Pramipexol Immediate Release
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexol Extended Release
  Arms: Pramipexole ER
Drug: Pramipexol Immediate Release
  Arms: Pramipexole IR
Drug: Placebo
  Arms: Placebo

SUMMARY:
The general aim of this trial is to determine the efficacy (as measured by the change from baseline to the end of the maintenance phase in the total score for Unified Parkinsons Disease Rating Scale Parts II and III combined), safety, and tolerability of pramipexole ER, in daily doses from 0.375 milligram to 4.5 milligram once a day, in comparison to placebo, in Levodopa combined with a Dopa-Decarboxylase-inhibitor treated Parkinson patients with advanced Parkinsons Disease and motor fluctuations.

In addition, a numerical comparison of the efficacy of pramipexole extended release versus pramipexole immediate release will be done.

The efficacy of pramipexole immediate release will also be compared to placebo, for assay sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with advanced idiopathic Parkinsons disease confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity.
2. Parkinsons disease diagnosed for at least 2 years.
3. Patients 30 years of age or older at the time of diagnosis.
4. Modified Hoehn and Yahr stage of 2 to 4 at on-time.
5. Treatment with standard or controlled release Levodopa combined with a Dopa-Decarboxylase-inhibitor, or with Levodopa combined with a Dopa-Decarboxylase-inhibitor/entacapone, at an optimised dose according to investigators judgement, this dose being stable for at least 4 weeks prior to baseline visit.
6. Motor fluctuations, with at least 2 cumulative hours of off-time every day during waking hours (documented on a patient diary completed for 2 consecutive days before baseline visit).
7. Patient willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures. In particular, after training, it has to be documented at baseline visit that the patient is able to recognise the off-time and on-time periods during waking hours and that the patient (or a family member or a guardian) is able to record them accurately in the patient diary.
8. Signed informed consent obtained before any study procedures are carried out (in accordance with International Conference on Harmonisation-Good Clinical Practice guidelines and local legislation).

Exclusion Criteria:

1. Atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis or degenerative diseases
2. Dementia, as defined by a Mini-Mental State Exam score < 24 at screening visit
3. Any psychiatric disorder according to Diagnostic and Statistical Manual of Mental Disorders 4th edition criteria that could prevent compliance or completion of the study and/or put the patient at risk if he/she takes part in the study
4. History of psychosis, except history of drug induced hallucinations
5. History of deep brain stimulation
6. Clinically significant Electrocardiogram abnormalities at screening visit
7. Clinically significant hypotension and/or symptomatic orthostatic hypotension at screening or baseline visit
8. Malignant melanoma or history of previously treated malignant melanoma
9. Any other clinically significant disease, whether treated or not, that could put the patient at risk or could prevent compliance or completion of the study
10. Pregnancy or breast-feeding
11. Sexually active female of childbearing potential not using a medically approved method of birth control for at least one month prior to the screening visit and throughout the study period
12. Serum levels of Aspartate Aminotransferase (Serum Glutamic-Oxaloacetic Transaminase), Alanine Aminotransferase (Serum Glutamic Pyruvic Transaminase), alkaline phosphatases or bilirubin > 2 Upper Limit of Normal
13. Patients with a creatinine clearance < 50 millilitres/minute
14. Any dopamine agonist (including pramipexole) within 4 weeks prior to baseline visit
15. Any medication with central dopaminergic antagonist activity within 4 weeks prior to the baseline visit
16. Any of the following drugs within 4 weeks prior to baseline visit: methylphenidate, cinnarizine, amphetamines
17. Flunarizine within 3 months prior to baseline visit
18. Known hypersensitivity to pramipexole or its excipients
19. Drug abuse according to investigators judgement, within 2 years prior to screening
20. Participation in other investigational drug studies, or use of other investigational drugs within one month or five times the half-life of the investigational drug (whichever is longer) prior to baseline visit

Min Age: 32 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (76):
- 248.525.43005 Boehringer Ingelheim Investigational Site, Linz, Austria
- Czechia (5):
  - 248.525.42003 Boehringer Ingelheim Investigational Site, Pardubice
  - 248.525.42001 Boehringer Ingelheim Investigational Site, Prague
  - 248.525.42005 Boehringer Ingelheim Investigational Site, Rakovník
  - 248.525.42002 Boehringer Ingelheim Investigational Site, Rychnov nad Kněžnou
  - 248.525.42004 Boehringer Ingelheim Investigational Site, Valašské Meziříčí
- Hungary (4):
  - 248.525.36005 Boehringer Ingelheim Investigational Site, Győr
  - 248.525.36003 Boehringer Ingelheim Investigational Site, Kecskemét
  - 248.525.36006 Boehringer Ingelheim Investigational Site, Szeged
  - 248.525.36004 Boehringer Ingelheim Investigational Site, Veszprém
- India (7):
  - 248.525.91004 National Institute of Mental Health & Neuro Sciences, Bangalore
  - 248.525.91002 Apollo Hospital, Chennai
  - 248.525.91001 Institute of Human Behaviour & Allied Sciences, Delhi
  - 248.525.91003 Nizam's Institute of Medical Sciences, Hyderabad
  - 248.525.91007 Boehringer Ingelheim Investigational Site, Indore
  - 248.525.91005 Mallikatta Neuro Research Center, Karnataka
  - 248.525.91006 King Edward Memorial Hospital & Research Centre, Pune
- Italy (8):
  - 248.525.39001 Policlinico di Catania, Catania
  - 248.525.39010 Campus Universitario Germaneto, Catanzaro
  - 248.525.39009 Ce.S.I., Chieti
  - 248.525.39007 Ospedale della Misericordia, Grosseto
  - 248.525.39002 Università Federico II, Napoli
  - 248.525.39008 Azienda Ospedaliera Pisana- Università degli Studi di Pisa, Pisa
  - 248.525.39005 Università La Sapienza di Roma, Roma
  - 248.525.39011 Policlinico Tor Vergata, Roma
- Philippines (8):
  - 248.525.63210 Makati Medical Center, Makati City
  - 248.525.63202 Chinese General Hospital, Manila
  - 248.525.63205 Jose Reyes Memorial Medical Center, Manila
  - 248.525.63206 Metropolitan Medical Center, Manila
  - 248.525.63207 Manila Doctors Hospital, Manila
  - 248.525.63201 The Medical City, Pasig
  - 248.525.63204 St Lukes Medical Center, Quezon
  - 248.525.63208 University of the East Ramon Magsaysay Memorial Medical Ctr, Quezon
- Poland (3):
  - 248.525.48001 Boehringer Ingelheim Investigational Site, Gdansk
  - 248.525.48003 Boehringer Ingelheim Investigational Site, Krakow
  - 248.525.48002 Wolski Hospital Dr. Anna Gostynska, Warsaw
- Russia (7):
  - 248.525.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 248.525.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 248.525.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 248.525.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 248.525.07007 Boehringer Ingelheim Investigational Site, Moscow
  - 248.525.07005 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 248.525.07006 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Slovakia (4):
  - 248.525.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 248.525.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 248.525.42103 Boehringer Ingelheim Investigational Site, Dubnica nad Váhom
  - 248.525.42101 Boehringer Ingelheim Investigational Site, Trnava
- South Korea (8):
  - 248.525.82001 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 248.525.82008 Boehringer Ingelheim Investigational Site, Kyeonggi-do
  - 248.525.82007 Boehringer Ingelheim Investigational Site, Pusan
  - 248.525.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 248.525.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 248.525.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 248.525.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 248.525.82006 Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - 248.525.34001 Boehringer Ingelheim Investigational Site, Alcorcon (Madrid)
  - 248.525.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 248.525.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 248.525.34005 Boehringer Ingelheim Investigational Site, Madrid
  - 248.525.34002 Boehringer Ingelheim Investigational Site, San Cugat Del Valles (Barcelona)
  - 248.525.34008 Boehringer Ingelheim Investigational Site, Tarrasa (Barcelona)
- Sweden (4):
  - 248.525.46005 Boehringer Ingelheim Investigational Site, Malmo
  - 248.525.46002 Boehringer Ingelheim Investigational Site, Nyköping
  - 248.525.46001 Boehringer Ingelheim Investigational Site, Stockholm
  - 248.525.46004 Boehringer Ingelheim Investigational Site, Stockholm
- Ukraine (6):
  - 248.525.38003 Boehringer Ingelheim Investigational Site, Dnipropetrovsk
  - 248.525.38006 Boehringer Ingelheim Investigational Site, Kharkiv
  - 248.525.38002 Boehringer Ingelheim Investigational Site, Kiev
  - 248.525.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 248.525.38001 Boehringer Ingelheim Investigational Site, Zaporizhzhya
  - 248.525.38005 Boehringer Ingelheim Investigational Site, Zaporizhzhya
- United Kingdom (5):
  - 248.525.44005 Boehringer Ingelheim Investigational Site, Barnsley
  - 248.525.44007 Boehringer Ingelheim Investigational Site, Blackburn
  - 248.525.44002 Boehringer Ingelheim Investigational Site, London
  - 248.525.44004 Boehringer Ingelheim Investigational Site, Norwich
  - 248.525.44003 Boehringer Ingelheim Investigational Site, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole ER: Pramipexole Extended Release (ER) (tablets of 0.375mg, 0.75mg, 1.5mg, 3.0mg or 4.5mg), dose: 0.375 mg, 0.75mg, 1.5mg, 2.25mg, 3.0mg, 3.75mg, or 4.5mg, mode of administration: Per os, once a day, in the morning
- Pramipexole IR: Pramipexole Immediate Release (IR) (tablets of 0.125mg, 0.25mg, 0.5mg, 1.0mg and 1.5mg), dose: 0.375mg, 0.75mg, 1.5mg, 2.25mg, 3.0mg, 3.75mg, or 4.5mg, mode of administration: Per os, in equally divided doses 3 times per day"
- Placebo: Matching Placebo to Pramipexole IR (tablets of 0.125mg, 0.25mg, 0.5mg, 1.0mg and 1.5mg), dose: 0.375mg, 0.75mg, 1.5mg, 2.25mg, 3.0mg, 3.75mg, or 4.5mg, mode of administration: Per os, in equally divided doses 3 times per day
  Matching Placebo to Pramipexole ER (tablets of 0.375mg, 0.75mg, 1.5mg, 3.0mg or 4.5mg), dose: 0.375 mg, 0.75mg, 1.5mg, 2.25mg, 3.0mg, 3.75mg, or 4.5mg, mode of administration: Per os, once a day, in the morning
Period: Overall Study
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Started | 165 | 175 | 178
Completed | 145 | 163 | 157
Not Completed | 20 | 12 | 21
Not completed — Adverse Event | 8 | 8 | 7
Not completed — Lack of Efficacy | 2 | 0 | 3
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 1 | 6
Not completed — patient did not meet inclusion criteria | 1 | 0 | 1
Not completed — Not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo | Total
Number analyzed (Participants) | 164 | 175 | 178 | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.7) | 62.0 (10.3) | 60.9 (9.7) | 61.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 77 | 84 | 233
  Male | 92 | 98 | 94 | 284

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Parts II+III Score at Week 18
Description: UPDRS II+III total score on Full Analysis Set (FAS)with LOCF (Last observation carried forward), week 18 - baseline, UPDRS II+III ranging from 0 (normal) to 160 (severe). UPDRS part II measures activities of daily living, part III measures motor symptoms
Time Frame: baseline and week 18
Population: Full analysis set (FAS 1) population = 507 patients FAS 1 defined as all patients who were dispensed study medication, were documented to have at least one dose of study medication, were treated for 18 weeks (or had prematurely discontinued treatment prior to week 18) and provided baseline and any on-drug post-baseline efficacy assessment
Measure: Least Squares Mean (Standard Error); unit: Percentage of change from baseline
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 161 | 172 | 174
Percentage of change from baseline | -11.0 (1.0) | -12.8 (0.9) | -6.1 (0.9)
Statistical Analysis 1: Comparison: Pramipexole ER vs Placebo; ANCOVA with factors treatment, pooled country and covariate baseline; Test type: Superiority or Other; p = 0.0001, ANCOVA; Adjusted mean difference from placebo = 4.9, 95% CI 2-sided [2.4 to 7.4], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Pramipexole IR vs Placebo; ANCOVA with factors treatment, pooled country and covariate baseline; Test type: Superiority or Other; p < .0001, ANCOVA; Adjusted mean difference from placebo = 6.6, 95% CI 2-sided [4.2 to 9.1], Standard Error of Mean 1.2

2. Secondary Outcome: Change From Baseline in Percentage Off-time at Week 18
Description: Percentage off-time based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). Off-time describes a period when the patient experiences increased parkinsonian symptoms (e.g. immobility or inability to move with ease).
Time Frame: baseline and week 18
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percentage of off-time
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 171 | 174
Percentage of off-time | -13.3 (1.4) | -15.9 (1.3) | -8.8 (1.3)
Statistical Analysis 1: Comparison: Pramipexole ER vs Placebo; ANCOVA with factors treatment, pooled country and covariate baseline; Test type: Superiority or Other; p = 0.0122, ANCOVA; Adjusted mean difference from Placebo = 4.5, 95% CI 2-sided [1.0 to 7.9], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: Pramipexole IR vs Placebo; ANCOVA with factors treatment, pooled country and covariate baseline; Test type: Superiority or Other; p < .0001, ANCOVA; Adjusted mean difference from placebo = 7.1, 95% CI 2-sided [3.7 to 10.5], Standard Error of Mean 1.7

3. Secondary Outcome: Change From Baseline in Percentage On-time Without Dyskinesia at Week 18
Description: Percentage on-time based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and week 18
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time without dyskinesia
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 171 | 174
Percentage of on-time without dyskinesia | 11.9 (1.7) | 12.6 (1.7) | 8.9 (1.6)

4. Secondary Outcome: Change From Baseline in Percentage On-time With Non-troublesome Dyskinesia at Week 18
Description: Percentage on-time with non-troublesome dyskinesia based on patient diary data, percentage ranging from 0 (worst case) to 100 (best case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and week 18
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 171 | 174
Percentage of on-time | 1.9 (1.2) | 3.9 (1.2) | 1.0 (1.2)

5. Secondary Outcome: Change From Baseline in Percentage On-time With Troublesome Dyskinesia at Week 18
Description: Percentage on-time with troublesome dyskinesia based on patient diary data, percentage ranging from 0 (best case) to 100 (worst case). On-time describes a period when the patient has no symptoms of off-time and is not asleep.
Time Frame: baseline and week 18
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Percentage of on-time
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 171 | 174
Percentage of on-time | -0.8 (0.5) | -0.8 (0.5) | -1.0 (0.5)

6. Secondary Outcome: Clinical Global Impression - Global Improvement (CGI-I) Responder
Description: CGI-I scores ranging from '1' (very much improved) to '7' (very much worse), CGI-I responder have scoring of 1 or 2 (at least much improved)
Time Frame: after 18 weeks of treatment
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 169 | 171
Participants
  Responder | 78 | 88 | 56
  Non-Responder | 82 | 81 | 115

7. Secondary Outcome: Response in Patient Global Impression (PGI-I)
Description: PGI-I scores ranging from '1' (very much better) to '7' (very much worse), PGI-I responder have scoring 1 or 2 (at least much better)
Time Frame: after 18 weeks of treatment
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 161 | 172 | 174
Participants
  Responder | 60 | 76 | 47
  Non-Responder | 101 | 96 | 127

8. Secondary Outcome: Change From Baseline in UPDRS I Score After 18 Weeks
Description: UPDRS I ranging from 0 (normal) to 16 (severe). UPDRS I measures Mentation, Behavior and Mood
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 161 | 172 | 174
Units on a scale | 0 [-1.0 to 0.0] | 0 [-1.0 to 0.0] | 0 [-1.0 to 0.0]

9. Secondary Outcome: Change From Baseline in UPDRS II Score After 18 Weeks, Average at on and Off-period
Description: UPDRS II ranging from 0 (normal) to 52 (severe). UPDRS Part II is calculated as the average of UPDRS part II at on and UPDRS part II at off-period for each of the 13 activities.
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 161 | 172 | 174
Units on a scale | -2.7 (0.3) | -3.6 (0.3) | -1.9 (0.3)

10. Secondary Outcome: Change From Baseline in UPDRS III Score After 18 Weeks
Description: UPDRS III ranging from 0 (normal) to 108 (severe). UPDRS part III measures motor symptoms
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 161 | 172 | 174
Units on a scale | -8.3 (0.7) | -9.2 (0.7) | -4.3 (0.7)

11. Secondary Outcome: Change From Baseline in UPDRS IV Score After 18 Weeks
Description: UPDRS IV ranging from 0 (normal) to 23 (severe). UPDRS IV measures complications of therapy
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 161 | 172 | 174
Units on a scale | -0.8 (0.2) | -0.9 (0.2) | -0.6 (0.2)

12. Secondary Outcome: Change From Baseline in Beck's Depression Inventory (BDI) After 18 Weeks
Description: ranging from 0 (best case) to 63 (worst case)
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 169 | 171
Units on a scale | -3.2 (0.5) | -4.0 (0.5) | -2.8 (0.5)

13. Secondary Outcome: Change From Baseline in Parkinson's Disease Sleep Scale (PDSS) After 18 Weeks
Description: ranging from 0 (worst case) to 150 (best case)
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 169 | 171
Units on a scale | 8.1 (1.8) | 8.9 (1.7) | 4.9 (1.7)

14. Secondary Outcome: Change From Baseline in Parkinson's Disease Quality of Life Questionnaire 39 After 18 Weeks
Description: Ranging from 0 (best case) to 156 (worst case)
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 149 | 165 | 164
Units on a scale | -9.1 (1.9) | -13.1 (1.8) | -6.2 (1.8)

15. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol) Scale After 18 Weeks
Description: ranging from 0 (worst case) to 100 (best case)
Time Frame: baseline and 18 weeks
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 150 | 165 | 164
Units on a scale | 5.8 (1.4) | 7.6 (1.3) | 4.3 (1.3)

16. Secondary Outcome: Change From Baseline in 11-point Likert Scale for Pain Related to PD at Week 18
Description: Likert scale is a method used for the measurement of pain. The patients were asked to rate their pain related to PD by ticking the number that best described their pain on the average in the previous week, from zero for "no pain" to ten for "unbearable pain".
Time Frame: baseline and week 18
Population: Full analysis set (FAS 1) population with last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 160 | 169 | 171
units on a scale | -0.4 (0.2) | -1.0 (0.2) | -0.3 (0.2)

17. Secondary Outcome: Clinically Significant Abnormalities: Clinical Laboratory Evaluations (Biochemistry and Haematology)
Time Frame: baseline and week 18
Population: Treated set (TS 1) population: defined as all patients who were dispensed study medication, were documented to have at least one dose of study medication and were treated for 18 weeks (or had discontinued treatment prior to week 18). Data limited to visit 8 (or V11 in case of premature discontinuation before visit 8).
Measure: Number; unit: participants
Arm/Group | Pramipexole ER | Pramipexole IR | Placebo
Number analyzed (Participants) | 150 | 162 | 158
participants
  Haematocrit - decrease | 2 [26.8 to 43.5] | 3 [32.4 to 48.8] | 1 [13.5 to 26.9]
  Haemoglobin - decrease | 2 | 5 | 3
  Red blood cell ct - decrease | 1 | 0 | 1
  Eosinophils - Increase | 3 | 2 | 1
  Neut.,poly. (segs),absol. - decrease | 0 | 1 | 0
  Sodium - decrease | 0 | 2 | 0
  GGT - increase | 1 | 0 | 1
  Glucose - decrease | 1 | 0 | 1
  Glucose - increase | 0 | 2 | 1
  Triglyceride - increase | 2 | 3 | 5
  Weight - decrease | 0 | 3 | 1
  Blood pressure - increase | 1 | 2 | 0
  Blood pressure - decrease | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of trial medication onwards up to the end of the trial (up to 34 weeks)
Description: After a 7-week double-blind flexible up-titration phase, there was an up to 26-week double-blind maintenance phase, followed by a 1-week downtitration phase (only for those patients not entering the open-label extension study).
Arm/Group | Placebo | Pramipexole ER | Pramipexole IR
Serious Adverse Events (participants affected / at risk) | 15/178 | 8/164 | 11/175
Other Adverse Events (participants affected / at risk) | 74/178 | 73/164 | 90/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=178) | Pramipexole ER (N=164) | Pramipexole IR (N=175)
Bronchitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Post viral fatigue syndrome (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Delusion (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
On and off phenomenon (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Radiculpathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Medical device change (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=178) | Pramipexole ER (N=164) | Pramipexole IR (N=175)
Nasopharyngitis (Infections and infestations) | 12 | 3 | 7
Anorexia (Metabolism and nutrition disorders) | 4 | 9 | 2
Hallucination (Psychiatric disorders) | 2 | 9 | 10
Insomnia (Psychiatric disorders) | 4 | 9 | 6
Dyskinesia (Nervous system disorders) | 16 | 28 | 34
Somnolence (Nervous system disorders) | 29 | 24 | 30
Dizziness (Nervous system disorders) | 9 | 9 | 19
Headache (Nervous system disorders) | 5 | 14 | 9
Nausea (Gastrointestinal disorders) | 19 | 18 | 20
Constipation (Gastrointestinal disorders) | 9 | 11 | 10
Vomiting (Gastrointestinal disorders) | 5 | 2 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.